CLINICAL TRIAL: NCT00179517
Title: Comparison of Anastrozole and Testosterone Versus Placebo and Testosterone Treatment of Reproductive and Sexual Dysfunction in Men With Epilepsy and Hypogonadism
Brief Title: Treatment of Sexual Dysfunction in Hypogonadal Men With Epilepsy With Testosterone and Either Anastrozole or Placebo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Andrew Herzog, Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2001P000149; IRUSANAS0004
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2017-08-08 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Seizure Disorder; Hypogonadism; Erectile Dysfunction
Keywords: Seizure; Epilepsy; Testosterone; Hormone; Sexual Dysfunction; Hypogonadism; Men
MeSH Terms: conditions — Epilepsy; Hypogonadism; Erectile Dysfunction; Seizures; Sexual Dysfunction, Physiological; Multiple Endocrine Neoplasia Type 1 | interventions — Anastrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- depotestosterone plus anastrozole (T-A) (Experimental): Each participant has biweekly intramuscular injections of 300 mg depotestosterone cypionate and takes an oral tablet of anastrozole 1 mg daily for the duration of the study. This group is referred to as the depotestosterone plus anastrozole (T-A) group.
  Interventions: Drug: Anastrozole 1mg
- depotestosterone plus placebo (T-P) (Placebo Comparator): Each participant has biweekly intramuscular injections of 300 mg depotestosterone cypionate and takes 1 matching placebo oral tablet daily for the duration of the study. This group is referred to as the depotestosterone plus placebo (T-P) group.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Anastrozole 1mg
  Other Names: Arimidex
  Arms: depotestosterone plus anastrozole (T-A)
Drug: Placebo Oral Tablet
  Arms: depotestosterone plus placebo (T-P)

SUMMARY:
The purpose of this study is to determine if treatment using a medication (anastrozole/Arimidex), which lowers estrogen levels in the blood is better than placebo, a tablet that does not contain any active medication, when combined with testosterone replacement to treat reproductive and sexual dysfunction in men with epilepsy. Anastrozole, the medication that is currently under study, does not, at this time, have FDA approval for use for this indication.

DETAILED DESCRIPTION:
This is a three-month study where baseline information is collected at the first visit and then each patient is started on treatment with testosterone supplementation and either anastrozole or placebo. Lab tests, seizure frequency, sexual function and mood will be monitored on a monthly basis.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a male between the ages of 18 and 50 years.
* Subject must have localization-related epilepsy with complex partial and/or secondary generalized seizures.
* Subject will meet criteria for hypogonadism (abnormally low bioactive testosterone levels and abnormally low scores on questionnaires of reproductive and sexual function).
* Subject will have had a normal urogenital and rectal/prostate exam during the year prior to entry.
* Subject will have had documentation of therapeutic range serum AED levels, a normal CBC, and hepatic enzyme (ALT,AST, alkaline phosphatase) levels that are less than twofold elevated during the 6 months prior to entry.

Exclusion Criteria:

* Subject that has taken hormones, major tranquilizers or antidepressants in the three months prior to entry.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2001-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Herzog, M.D., M.Sc., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herzog AG, Farina EL, Drislane FW, Schomer DL, Smithson SD, Fowler KM, Dworetzky BA, Bromfield EB. A comparison of anastrozole and testosterone versus placebo and testosterone for treatment of sexual dysfunction in men with epilepsy and hypogonadism. Epilepsy Behav. 2010 Feb;17(2):264-71. doi: 10.1016/j.yebeh.2009.12.003. Epub 2010 Jan 21. PMID 20096638

RESULTS

PARTICIPANT FLOW:
Groups:
- Depotestosterone Plus Anastrozole (T-A): Each participant has biweekly intramuscular injections of 300 mg depotestosterone cypionate and takes 1 mg of anastrozole daily for the duration of the study.
  Anastrozole 1mg
- Depotestosterone Plus Placebo (T-P): Each participant has biweekly intramuscular injections of 300 mg depotestosterone cypionate and takes 1 matching placebo tablet daily for the duration of the study.
  Placebo Oral Tablet
Period: Overall Study
Arm/Group | Depotestosterone Plus Anastrozole (T-A) | Depotestosterone Plus Placebo (T-P)
Started | 20 | 20
Completed | 18 | 19
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Depotestosterone Plus Anastrozole (T-A) | Depotestosterone Plus Placebo (T-P) | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (7.5) | 42.7 (7.2) | 43.0 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 19 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 19 | 37
Participants with Epilepsy [Count of Participants; unit: Participants] | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Sexual Function Scores, Calculated Using S-Score and Reynolds' Sexual Questionnaires, Will Increase More Anastrozole and Testosterone Treatment Than With Placebo and Testosterone Treatment.
Description: S-Scores and Reynolds Questionnaire scores were assessed at baseline and once a month over three months. The average change in score for each questionnaire over the 3 month study was reported. The S-Scores questionnaire measured sexual function and consisted of four questions with five possible answers. The total scale range was 0-20, with higher scores were considered better. S-Scores that were greater than or equal to 16/20 were considered normalized S-Scores. Reynolds Questionnaire is a 21 item survey that monitors sexual interest, activity, satisfaction, and function. The scale for the Reynolds questionnaire for sexual interest was from 0-12, with higher scores being better. The scale for sexual activity was 0-41 with higher scores being better. The sexual satisfaction scale was from 0-21 with higher scores being better. The scale for sexual function was from 0 to -12 with lower scores being better.
Time Frame: 3 month average
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Depotestosterone Plus Anastrozole (T-A) | Depotestosterone Plus Placebo (T-P)
Number analyzed (Participants) | 18 | 19
Scores on a Scale
  Change in S-Score | 3.7 (1.6) | 2.5 (2.2)
  Reynolds Questionnaire Change in R-Interest | 2.4 (2.1) | 1.5 (2.6)
  Reynolds Questionnaire Change in R-Activity | 11.1 (25.7) | 4.7 (7.9)
  Reynolds Questionnaire Change in R-Satisfaction | 2.4 (3.7) | 2.1 (3.3)
  Reynolds Questionnaire Change in R-Function | -1.7 (7.4) | -1.3 (4.1)

2. Secondary Outcome: The Proportion of Men Who Achieve Normalization of Sexual Scores (Sexual Interest Function,) Using Anastrozole and Placebo
Description: The proportion of men who achieve normalization of sexual scores (scores greater than or equal to 16/20) on anastrozole (T-A) and those on placebo (T-P) are reported. Both Men who achieve normalization of sexual scores and those who did not achieve normalization of sexual scores were reported for anastrozole (T-A) treatment group and the placebo treatment group. Sexual scores were gathered once per month for three months with the average of the three months reported.
Time Frame: Assessed for 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Depotestosterone Plus Anastrozole (T-A) | Depotestosterone Plus Placebo (T-P)
Number analyzed (Participants) | 18 | 19
Participants
  Normalization of S-Score | 13 | 9
  No Normalization of S-Score | 5 | 10

3. Secondary Outcome: Bioavailable Testosterone Levels in Subjects on Anastrozole (T-A) and Subjects on Placebo (T-P).
Description: Bioavailable testosterone levels were measured at baseline and once a month over the three month study. The average change in bioactive testosterone levels from baseline to the end of the three month study was reported.
Time Frame: Assessed for 3 months
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Depotestosterone Plus Anastrozole (T-A) | Depotestosterone Plus Placebo (T-P)
Number analyzed (Participants) | 18 | 19
ng/dl | 150.9 (144.0) | 161.7 (123.1)

4. Secondary Outcome: Estradiol Levels in Subjects on Anastrozole (T-A) and Subjects on Placebo (T-P).
Description: Estradiol levels were measured once a month over the three month study in subjects taking anastrozole (T-A) and in subjects taking placebo (T-P). The average change in estradiol levels was reported.
Time Frame: Assessed for 3 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Depotestosterone Plus Anastrozole (T-A) | Depotestosterone Plus Placebo (T-P)
Number analyzed (Participants) | 18 | 19
pg/mL | -14.6 (17.3) | 8.6 (19.6)

5. Secondary Outcome: The Bioavailable Testosterone and Estradiol Ratio in Subjects Taking Anastrozole and Subjects Taking Placebo.
Description: Bioavailable testosterone and estradiol levels were measured once a month over the three month study in subjects taking anastrozole and subjects taking placebo. The bioavailable testosterone and estradiol levels for the three months were averaged for each subject. The ratio between the average bioavailable testosterone level and average estradiol levels were reported.
Time Frame: Assessed for 3 months
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Depotestosterone Plus Anastrozole (T-A) | Depotestosterone Plus Placebo (T-P)
Number analyzed (Participants) | 18 | 19
Ratio | 145.47 (143.00) | 12.78 (10.21)

6. Secondary Outcome: Bioavailable Testosterone and Luteinizing Hormone Ratios in Subjects Taking Anastrozole (T-A) and in Subjects Taking Placebo (T-P).
Description: Bioavailable Testosterone and luteinizing hormone levels were measured once a month over the three month study in the treatment and placebo group. The bioactive testosterone and luteinizing hormone levels were averaged for the three months. The ratio between the average bioactive testosterone level and average luteinizing hormone levels were reported.
Time Frame: Assessed for 3 months
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Depotestosterone Plus Anastrozole (T-A) | Depotestosterone Plus Placebo (T-P)
Number analyzed (Participants) | 18 | 19
Ratio | 450.24 (193.17) | 482.65 (346.10)

7. Secondary Outcome: Estradiol and Luteinizing Hormone Ratios in Subjects Taking Anastrozole (T-A) and in Subjects Taking Placebo (T-P).
Description: Estradiol and luteinizing hormone levels were measured once a month over the three month study in the treatment and placebo group. The estradiol and luteinizing hormone levels were averaged for the three months. The ratio between the average estradiol levels and average luteinizing hormone levels were reported.
Time Frame: Assessed for 3 months
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Depotestosterone Plus Anastrozole (T-A) | Depotestosterone Plus Placebo (T-P)
Number analyzed (Participants) | 18 | 19
Ratio | 9.31 (8.84) | 53.80 (47.25)

8. Secondary Outcome: Changes in Seizure Frequency in Subjects Taking Anastrozole (T-A) and Subjects Taking Placebo (T-P).
Description: The average change in number of seizures over the 3 month study for the depotestosterone plus anastrozole (T-A) and depotestosterone plus placebo (T-P) were reported.
Time Frame: Assessed for 3 months
Measure: Mean (Standard Deviation); unit: number of seizures
Arm/Group | Depotestosterone Plus Anastrozole (T-A) | Depotestosterone Plus Placebo (T-P)
Number analyzed (Participants) | 18 | 19
number of seizures | -2.0 (1.2) | -2.9 (2.9)

9. Secondary Outcome: Changes in Energy, Mood and Anxiety Scores for Subjects Taking Anastrozole (T-A) and for Subjects Taking Placebo (T-P).
Description: Changes in energy, mood and anxiety scores were measured using The Beck Depression Inventory II and the POMS questionnaire. The Beck Depression Inventory II questionnaire consisted of 21 questions, each with answers ranging from 0-3. The answers for each question were summed. The scale ranged from 0-63 with higher scores meaning a higher depression score (worse score). The POMS questionnaire had a total of 65 questions that measured tension, depression, anger, vigor, fatigue and confusion. The total POMS score ranged from 0-200, with lower scores being better. The POMS tension score ranged from 0-36 with lower scores being better. The POMS depression score ranged from 0-60 with lower scores being better. The POMS anger score ranged from 0-48, lower scores being better. The POMS vigor score ranged from 0-32, lower scores being better. The POMS fatigue score ranged from 0-28, lower scores being better. The POMS confusion score ranged from 0-28 with lower scores being better.
Time Frame: Assessed for 3 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Depotestosterone Plus Anastrozole (T-A) | Depotestosterone Plus Placebo (T-P)
Number analyzed (Participants) | 18 | 19
Scores on a scale
  Change in Depression (Beck Depression Inventory II | -5.3 (7.6) | -6.4 (9.4)
  Change in Vigor | 4.6 (5.9) | 4.8 (7.6)
  Change in Fatigue | -6.0 (5.4) | -4.5 (8.1)
  Change in Depression (POMS-D) | -5.6 (0.6) | -6.7 (11.5)
  Change in Anxiety (POMS-T) | -3.0 (5.8) | -4.2 (7.4)
  Change in Anger (POMS A) | -2.4 (8.7) | -2.6 (8.9)
  Change in Confusion (POMS-C) | -2.7 (4.1) | -2.7 (5.7)

ADVERSE EVENTS:
Arm/Group | Depotestosterone Plus Anastrozole (T-A) | Depotestosterone Plus Placebo (T-P)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 0/18 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No